CLINICAL TRIAL: NCT03424538
Title: The Effect of Variable Intensity Work on Postural Instability, Motion Performance and Quality of Life in Multiple Sclerosis Patients
Brief Title: The Effect of Neurorehabilitation Therapy on Postural Control, Mobility and Quality of Life in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Tollár József, Principal Investigator, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB008/2017
Record Dates: First submitted 2018-01-18; First posted 2018-02-07 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2018-03

CONDITIONS: Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Primary Progressive
Keywords: multiple sclerosis; posture; neurorehabilitation; balance
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Neurological Rehabilitation; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: The single-arm, 5-week intervention is monitor every day on the effect of postural control on walking performance, balance and quality of life. The intervention team (n = 15) takes 25 training sessions for 5 weeks. Every move takes 60 minutes to continuously increase the load intensity of the X-box program. Before each intervention started, the patients perform a 10 minute warm-up and the drainage exercises are 15 minutes stretching exercises. The MStp group (n=14) participated in a 5-week physiotherapy course. The general treatment consisted of strengthening, stretching and walking correction. During the 5-week period, 25 patients attended training. One treatment takes 60 minutes. The control group (n = 14) did not receive physiotherapeutic treatment outside the medication.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MSt (Experimental): The MSt group that received 5 weeks of intensive therapy.
  Interventions: Other: Neurorehabilitation
- MSc (No Intervention): The MS controll group that did not receive treatment.
- MStp (Experimental): The MStp Group performs a traditional physiotherapy for 5 weeks.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Neurorehabilitation — 5-week-long intervention, administered daily, targeted postural instability, balance and mobility using at-limit intensity sensorimotor and visuomotor agility training
  Arms: MSt
Other: Physiotherapy — 5-week-long intervention, physiotherapy, stretching, walking preparation, strengthening
  Arms: MStp

SUMMARY:
Abstract Introduction: Postural control disorders are the most common motor disorder associated with multiple sclerosis.

Objective: The aim of this study is to demonstrate the potential for improvement of postural control, motion performance and quality of life in patients with multiple sclerosis who are performing a special neurorevolutionary balancing program.

Intervention: The treated group (n = 15) performed five times a week for the treatment we defined. (60 minutes per day). The experimental group performed movements using the Xbox 360 and Kinect consoles. The study team participated in 25 sessions, five times a week. The duration of treatment was 5 weeks.The MStp group (n=14) participated in a 5-week physiotherapy course. The general treatment consisted of strengthening, stretching and walking correction. During the 5-week period, 25 patients attended training. One treatment takes 60 minutes. Sensory Organisation Test / Body Sway at the end of the baseline and treatment protocol is used to evaluate each patient. The quality of life mapping was measured by subjective tests (EQ-5D-5L, ADL). To assess the depressive state, a Beck depression questionnaire was used. Balance and motion performance were used by the Berg Balance Test and 6Minutes Walk Test. The results were compared with the control group results (n = 14) and showed improvement in overall balance and motion performance.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis
* instability problem

Exclusion Criteria:

* Severe heart problems, severe demeanor, alcoholism, drug problems

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
Postural instability | 5 weeks
  Body sway (mm) (Posturography test)
quality of life | 5 weeks
  EQ-5D (EQ-5D was first introduced in 1990 by the EuroQol Group, The EQ-5D questionnaire is made up for two components; health state description and evaluation)
balance test | 5 weeks
  Berg Balance test (The Berg Balance Scale (BBS) was developed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks, 41-56 = low fall risk, 21-40 = medium fall risk, 0 -20 = high fall risk )
mobility test | 5 weeks
  Six minutes walk test (6MWT) (m) (The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway)

SECONDARY OUTCOMES:
depression scale | 5 weeks
  Beck Depression scale (The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression, 0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, 29-63: severe depression)

CONTACTS AND LOCATIONS:
Overall Officials: József Tollár, MSC, Principal Investigator — Somogy Megyei Kaposi Mór Teaching Hospital
Locations (1):
- Somogy Megyei Kaposi Mór Teaching Hospital, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: description related info — https://www.ncbi.nlm.nih.gov/pubmed/?term=multiple+sclerosis+rehabilitation+wii